CLINICAL TRIAL: NCT00704418
Title: Efficacy and Safety of Bromfenac Ophthalmic Solution in Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-S&E-0415081-P-WR
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Results first posted 2011-01-26 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Cataract
Keywords: Cataract extraction; intraocular lens implantation
MeSH Terms: conditions — Cataract | interventions — bromfenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bromfenac (Experimental): Bromfenac ophthalmic solution 0.09%, dosed 1 drop daily
  Interventions: Drug: Bromfenac
- Placebo (Placebo Comparator): Placebo, dosed 1 drop daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bromfenac — sterile ophthalmic solution
  Arms: Bromfenac
Drug: Placebo — sterile ophthalmic solution
  Arms: Placebo

SUMMARY:
Efficacy and Safety of Bromfenac Ophthalmic Solution in Cataract Surgery

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for cataract surgery

Exclusion Criteria:

* Known hypersensitivity to bromfenac and salicylates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ISTA Pharmaceuticals, Inc., Irvine, California, United States

REFERENCES:
- [Derived] Silverstein SM, Cable MG, Sadri E, Peace JH, Fong R, Chandler SP, Gow JA, Klier SM, McNamara TR; Bromfenac Ophthalmic Solution Once Daily (Bromday) Study Group. Once daily dosing of bromfenac ophthalmic solution 0.09% for postoperative ocular inflammation and pain. Curr Med Res Opin. 2011 Sep;27(9):1693-703. doi: 10.1185/03007995.2011.597663. Epub 2011 Jul 14. PMID 21751945

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 19 sites, first participant entered the study 06/03/2008 and last participant completed the study 08/29/2008.
Pre-assignment Details: A total of 156 participants were randomized to investigational product and were included in the Intent-to-Treat (ITT) population; 78 were randomized to the bromfenac ophthalmic solution treatment group and 78 were randomized to the placebo treatment group.
Period: Overall Study
Arm/Group | Bromfenac | Placebo
Started | 78 | 78
Completed | 73 | 72
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Over-enrolled/surgery postponed | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bromfenac | Placebo | Total
Number analyzed (Participants) | 78 | 78 | 156
Age Continuous [Mean (Full Range); unit: years] | 68.7 [27.0 to 90.0] | 68.0 [43.0 to 86.0] | 68.4 [27.0 to 90.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 48 | 93
  Male | 33 | 30 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Summed Ocular Inflammation Score (SOIS) of Zero
Description: Participants with SOIS of 0. Scale: 0=0 cells (complete absence); 0.5=1-5 cells; 1=6-15 cells (very slight); 2=16-25 cells (moderate); 3=26-50 cells (marked); 4=>50 cells (intense)
Time Frame: Day 15
Population: Last Observation Carried Forward Analysis(LOCF), ITT Population
Measure: Number; unit: participants
Arm/Group | Bromfenac | Placebo
Number analyzed (Participants) | 78 | 78
participants | 36 | 23

2. Secondary Outcome: Number of Participants That Are Pain Free
Description: Participant description of being pain free (Score of none)taken from patient questionnaire, Ocular Comfort Grading Assessment with multiple possible responses
Time Frame: Day 1
Population: LOCF Analysis, ITT Population
Measure: Number; unit: participants
Arm/Group | Bromfenac | Placebo
Number analyzed (Participants) | 78 | 77
participants | 65 | 40

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Bromfenac | Placebo
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/73
Other Adverse Events (participants affected / at risk) | 6/73 | 19/73
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bromfenac (N=73) | Placebo (N=73)
Corneal oedema (Eye disorders) | 0 (0) | 4 (5)
Eye Pain (Eye disorders) | 2 (2) | 5 (5)
Eye Inflammation (Eye disorders) | 4 (5) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the PI will provide to the sponsor a copy of proposed publication information for review, comment and approval following completion of the study and at least sixty (60) days prior to submission of the publication. If sponsor requests in writing, the PI will withhold publication until written permission is given by sponsor.